CLINICAL TRIAL: NCT06726538
Title: Investigating the Efficacy of Autologous, Adipose-derived Mesenchymal Stem Cell Therapy in Women Aged 40-50
Brief Title: Investigating the Efficacy of Autologous, Adipose-derived Mesenchymal Stem Cell Therapy for the Treatment of Sexual Function Impairment in Women Aged 40-50
Acronym: IEAAMSC-W40-50
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vinmec Research Institute of Stem Cell and Gene Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISC.01230086
Record Dates: First submitted 2024-12-02; First posted 2024-12-10 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Female Sexual Dysfunction
Keywords: female sexual dysfunction; sexual function impairment; adipose-derived mesenchymal stem cell therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSC infusion group (Group A) (Experimental): This clinical trial involves intravenous administration of MSCs at a dose of 10^6 cells/kg, offering a non-rejection approach due to the autologous nature of the cells. These cells, surviving approximately 8 weeks in the body, secrete growth factors and cytokines to nourish cells, enhance vascular supply, and mitigate harmful inflammation, thereby countering cellular aging. Fifty female participants will be randomly assigned to two groups. Group A will receive mesenchymal stem cell (MSC) infusions twice: once at baseline and a second time three months later.
  Interventions: Biological: Intravenous administration of Autologous, adipose-derived mesenchymal stem cells
- Control group (Group B) (No Intervention): 25 participants in Group B will act as controls for 6 months.

INTERVENTIONS:
Biological: Intravenous administration of Autologous, adipose-derived mesenchymal stem cells — Patients in group A will receive two infusions of autologous, adipose-derived mesenchymal stem cells at day 0 and day 90 ± 14 at a dose of 10^6 cells/kg.
  Autologous, adipose-derived mesenchymal stem cells used in this study were harvested from autologous fat tissue through an enzyme method and expanded using our in-house optimized serum-free and xeno-free culture under a physiological oxygen concentration of 5%. For clinical use, cells at passage 3 will be harvested in 100 mL Ringer's lactate. Therapeutic ASC products must pass the following releasing criteria: (1) negative for bacteria, fungi and mycoplasma; (2) more than 90% viability; (3) expression of more than 95% positivity for CD105, CD73, and CD90 and less than 2% positivity for CD45, CD34, CD11b, CD19, and HLA-DR; and (4) endotoxin <5 EU/kg. The patient will be infused with 1x106 cells/kg body weight within 60 minutes via the intravenous route.
  Arms: MSC infusion group (Group A)

SUMMARY:
Female Sexual Dysfunction (FSD) represents a critical public health challenge, significantly impacting women's physical, psychological, and social well-being. Despite its prevalence, cultural barriers in Vietnam and other Asian countries often limit awareness and research on FSD. Existing treatments, such as hormone therapy, carry risks like cardiovascular complications and cancer, emphasizing the need for innovative interventions. This study investigates FSD-related factors and evaluates the efficacy of autologous adipose-derived mesenchymal stem cell (MSC) therapy as a novel approach.

In this phase 2 clinical trial, MSCs are intravenously administered at a dose of 10^6 cells/kg. These autologous cells, which are non-immunogenic, survive for approximately 8 weeks and release growth factors and cytokines to enhance vascular supply, reduce harmful inflammation, and counteract cellular aging. The study enrolls 50 female participants randomized into two groups: Group A receives MSC infusions at months 0 and 3, while Group B acts as a control for 6 months.

Outcomes are assessed through clinical evaluations, blood tests for hormonal levels, molecular analyses, and internationally validated quality-of-life and sexual function scales. Evaluations are conducted at baseline, 3, and 6 months post-infusion. This research seeks to provide robust evidence for the safety and efficacy of MSC therapy, offering a promising alternative to conventional treatments while addressing a critical gap in women's health.

DETAILED DESCRIPTION:
Female Sexual Dysfunction (FSD) is a significant public health concern. FSD can lead to various health issues and increase the risk of developing other conditions such as osteoporosis, cardiovascular diseases, and cancer. Although hormone therapy is commonly used to treat FSD, its long-term use may have adverse effects on cardiovascular health and raise the risk of cancer. Therefore, exploring new, safe, and effective treatment methods is essential. In 2015, the FDA approved the use of flibanserin (Addyi® Sprout Pharmaceuticals, USA) for premenopausal women with reduced sexual desire. However, this therapy remains controversial due to its potential side effects and limited efficacy. Current treatments for Female Sexual Dysfunction (FSD) mainly involve hormone replacement therapy, gonadotropin therapy, dietary supplements, or lifestyle modifications. While hormone therapy is commonly used to address hormonal decline in women, long-term use may lead to cardiovascular issues or cancer. Therefore, exploring psychological therapies and researching new potential treatments to meet patients' needs is essential.

Recent studies suggest that mesenchymal stem cells (MSCs) offer a safe approach to restoring hormone deficiencies. Clinical trials have investigated the use of MSC transplants to treat conditions like premature ovarian failure and ovarian cancer. Numerous trials have employed MSCs derived from bone marrow, umbilical cords, adipose tissue, or menstrual blood to address ovarian and uterine dysfunctions. Edessy et al. reported using autologous stem cells to treat 10 participants with premature ovarian failure. Following transplantation, two participants resumed menstruation within three months, one of whom became pregnant after 11 months and delivered a healthy full-term baby. Hormonal tests in the pregnant case revealed restored levels of FSH, LH, E2, and AMH to normal ranges. Although these studies are limited by small sample sizes and the lack of control groups, they highlight the potential of MSC transplantation as a treatment for FSD.

A study by Mashayekhi et al. demonstrated the safety of autologous adipose-derived mesenchymal stem cell (MSC) therapy for premature ovarian failure, with no adverse effects reported among nine participants receiving different cell doses. Menstruation resumed in two participants in both the high-dose (15x10^6 cells/kg) and lower-dose (5x10^6 and 10x10^6 cells/kg) groups, while serum FSH levels improved in four participants. Despite small sample size and lack of a control group, the study supports the safety of MSC infusion into the ovaries. Another ongoing trial (NCT01853501) aims to further investigate MSC therapy for ovarian failure, though results are pending. In Vietnam, the Vinmec Institute of Stem Cell and Gene Technology conducted a study on Female Sexual Dysfunction (FSD), using intravenous MSC infusions for 16 women. The trial reported no adverse effects, with participants reporting improved satisfaction with sexual health, though hormone levels (AMH, FSH, and E2) showed no significant changes.

This study aims to address the need for a novel and more effective approach to treating hormonal decline in women, not only improving sexual function but also enhancing their quality of life. Based on this rationale, we have decided to conduct the study titled "Investigating the efficacy of autologous, adipose-derived mesenchymal stem cell therapy for the treatment of sexual function impairment in women aged 40-50," with the following objective: Evaluate the improvement in sexual function among women aged 40-50 years who received autologous adipose-derived mesenchymal stem cell (MSC) therapy.

ELIGIBILITY:
Inclusion Criteria:

* Women between 40 - 50 years of age and have not gone through menopause
* The last menstrual period before participating in the study at least 2 months or more
* FSH before the menopause (tested on 2nd - 7th day of the menstrual cycle): FSH ≤ 29.8 mIU/mL
* FSFI < 26.55 ± signs of decline in sexual or reproductive functions such as symptoms of premenopausal such as hot flashes, excessive sweating, headaches
* Normal liver function
* Normal kidney function
* Normal cardiovascular function

Exclusion Criteria:

* Previous surgery to remove gonads
* Diagnosed with cancer
* Had an organ transplant
* Has congenital malformations related to the gonads
* Diagnosed with chronic diseases such as diabetes, hypopituitarism, adrenal insufficiency, and blood pressure unresponsive to treatment
* Diagnosis of active autoimmune diseases

Ages: 40 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study is open to individuals who self-identify as female. Participants must be biologically female and within the age range of the study criteria, as the research focuses on addressing Female Sexual Dysfunction (FSD) and related factors specific to women.
Enrollment: 50 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
The safety of autologous, adipose-derived mesenchymal stem cell therapy based on The number of adverse events (AEs) and serious adverse events (SAEs) | at baseline, 3, and 6 months post-infusion
  Adverse Events (AEs): refer to any unfavorable or unintended signs, symptoms, or diseases that occur in a participant during a study or treatment, regardless of whether they are causally related to the intervention.
  Serious Adverse Events (SAEs): Events are a subset of adverse events that meet specific criteria (e.g., hospitalization, life-threatening situations) indicating a higher level of severity.
Changes in sexual functions of participants based on the Female Sexual Function Index | at baseline, 3, and 6 months post-infusion
  based on the Self-Assessment Questionnaires: the Vietnamese versions of Female Sexual Function Index (FSFI). The Female Sexual Function Index (FSFI) is a 19-item questionnaire scored on a 5-point Likert scale, designed to assess six key domains of female sexual function: desire, arousal, lubrication, orgasm, satisfaction, and pain. Total scores range from 2 to 36, with higher scores indicating better sexual function, while scores below 26.55 suggest a risk of dysfunction.
Changes in sexual functions of participants based on the AMS Diagnosing Menopause | at baseline, 3, and 6 months post-infusion
  The Self-Assessment Questionnaires: the AMS Diagnosing Menopause (AMS): the severity of problem is scored as follows score: None =0; Mild =1; Moderate =2; Severe =3. The symptoms are grouped into 4 categories, vasomotor, psychological, locomotor and urogenital. A score of 15 or over usually indicates lower sexual function
Changes in sexual functions of participants based on the UTIAN Quality of Life Scale (UQOL) | at baseline, 3, and 6 months post-infusion
  The Utian QOL scale (UQOL) that is strongly based on perception of sense of well-being as distinct from menopausal symptoms. The UQOL contains 23 items divided into four domains: Occupational (7 items); Health (7 items); Emotional (6 items); Sexual (3 items). Total Score: 23-115. Higher scores indicate a better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Liem Thanh Nguyen, PhD, Study Director — Vinmec Research Insitute of Stem Cell and Gene Technology
Locations (2):
- Vietnam (2):
  - Vinmec Research Institute of Stem Cell and Gene Technology, Hanoi
  - Vinmec Times City International Hospital, Hanoi